CLINICAL TRIAL: NCT06920303
Title: Accuracy of Transcranial Colour Coded Duplex Compared With CT Angiography in Diagnosing Arterial Obstructions in Acute Ischemic Strokes
Brief Title: Accuracy of Transcranial Colour Coded Duplex in Comparing With CT Angiography
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hassan Hamdy Hamed, Resident-neurology and psychological medicine department-Sohag hospital university, Sohag University
Other Study IDs: Soh-Med--25-3-01MS
Record Dates: First submitted 2025-03-30; First posted 2025-04-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke, Acute
Keywords: transcranial colour coded duplex; ct angiography
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- patients who suffer from ischemic cerebrovascular stroke: All subjects must meet the following criteria to be enrolled in the study, patients who have ischemic strokes or transient ischemic attacks and will be admitted in department of neurology and psychological medicine and stroke unit at Sohag university hospital.
  Interventions: Device: transcranial colour coded duplex

INTERVENTIONS:
Device: transcranial colour coded duplex — transcranial colour coded duplex is good non invasive tool in detect velocity and obstructions of intracranial arteries

SUMMARY:
Investigator will compare accuracy of transcranial colour coded duplex with CT angiography in detecting arterial obstructions in patients presenting or with history of cerebrovascular ischemic strokes

DETAILED DESCRIPTION:
Cerebrovascular stroke is one of the most common causes of death and disability in the World. It accounts for almost 5% of all disability-adjusted life-years and 10% of all deaths worldwide.

Atherosclerosis is one of the major causes of ischemic stroke, it can lead to cerebrovascular stroke through progressive stenosis, occlusion of the extra or intracranial vessels and or arterio-arterial embolization from an atheromatous plaque.

Intracranial stenosis presents with one or recurrent ischemic strokes and transient ischemic attacks.

High-grade stenosis contributes to both the occurrence and magnitude of ischemic injury.

Overall, 50% of patients have either lacunar, subcortical, or cortical infarction.

The remaining patients with intracranial stenosis have multiple lesions involving a combination of cortical, subcortical, and lacunar infarctions.

There are extensive data about carotid atherosclerosis from American, European and Asian population. However, data from Egyptian ethnics are extremely rare.

Ethnic-racial factors are related to the development of extra- and intracranial atherosclerosis.

Intracranial stenosis causes about 10% of strokes in white people, 20-29% of transient ischemic attacks or strokes in black people, and up to 40-50% of strokes in Asian people.

Extracranial atherosclerosis is common among Caucasian stroke patients. For example, in the United States and Western communities, extracranial carotid artery disease was estimated to be responsible for 20-30% of strokes, while less common in Asian and African populations.

Intracranial arterial stenosis is prevalent in the Egyptian stroke population, similar to most non-white populations.

Transcranial Doppler is routinely performed to assess the blood flow in patients with cerebral ischaemia and provides important real-time information about cerebral haemodynamics.

Transcranial doppler can aid in the diagnostic work-up by detecting, localising and grading the severity of intracranial arterial obstruction.

Transcranial Doppler is an established tool for the non-invasive assessment of cerebral blood flow. Since transcranial doppler results vary with the skills and experience of the sonographer, it requires validation against contrast angiography.

ELIGIBILITY:
Inclusion Criteria:

* patients who have acute ischemic strokes or transient ischemic attacks .

Exclusion Criteria:

1. Patients with history of cardiac arrhythmia or discovered recently or known rheumatic heart disease.
2. Patients with history of autoimmune diseases.
3. Patients with space occupying lesion or hemorrhage in Ct brain.
4. Pregnant female.
5. Patients who refuse to participate in the study.
6. Patients who have history of allergy or developed acute kidney injury during previous dye injection.
7. Patients who have chronic kidney disease.
8. Premorbid neurological disorder (myopathy, multiple sclerosis) on neurological examination or previous investigations.
9. Inability to achieve safe vascular access.
10. Patients with insufficient temporal acoustic window.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: one hundred cases of patients with acute ischemiac cerebrovascular stroke will be included in the study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
detect accuracy of transcranial color coded duplex compared with CT angiography in diagnosing arterial obstructions in acute ischemic stroke | one year after enrolling one hundred cases
  investigator will detect if transcranial color coded duplex can be used for diagnosing arterial obstructions in acute ischemic stroke by measuring the peak systolic velocity of different intracranial arteries, investigator will compare with CT angiography imaging results to assess the accuracy of transcranial color coded duplex in diagnosis of acute ischemic stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. DALYs GBD, Collaborators H. Global, regional, and national disability-adjusted life-years (DALYs) for 359 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018;392(10159):1859-922. 2. Johansson BB. Hypertension mechanisms causing stroke. Clin Exp Pharmacol Physiol. 1999;26(7):563-5.. 3. Grau AJ, Weimar C, Buggle F, Heinrich A, Goertler M, Neumaier S, et al. Risk factors, outcome, and treatment in subtypes of ischemic stroke: the German stroke data bank. Stroke. 2001;32(11):2559-66.. 4. Meseguer E, Lavallee PC, Mazighi M, et al. Yield of systematic transcranial Doppler in patients with transient ischemic attack. Ann Neurol 2010;68:9-17.